CLINICAL TRIAL: NCT04701398
Title: Frailty in Patients With Advanced Chronic Kidney Disease Waiting for a Kidney Transplantation. A Randomized Clinical Trial of Multimodal Prehabilitation.
Brief Title: Multimodal Prehabilitation in Frail and Non-frail Patients Waiting for a Kidney Transplantation (the FRAILMAR Study)
Acronym: Frailmar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI19/0037
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; kidney transplantation; frailty; prehabilitation; exercise; nutritional status; psychological advice; sarcopenia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Frailty; Motor Activity; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal intervention (Experimental): supervised physical training (1-hour sessions, 24 sessions, 8 weeks) + nutritional supplementation + psychological advice
  Interventions: Other: Multimodal prehabilitation
- Standard Care (No Intervention): Healthy living recommendations

INTERVENTIONS:
Other: Multimodal prehabilitation — Exercise + nutritional supplementation + psychological advice
  Arms: Multimodal intervention

SUMMARY:
Frailty is very frequent among patients waiting for a kidney transplantation (KT). Frailty and poor fitness powerfully predict mortality, kidney graft survival, and healthcare utilization after KT. Frailty in patients with chronic kidney disease (CKD) displays a constellation of features that characterize a special population. Intervention is essential to improve quality of life for frail CKD patients, regardless of their age. A pre-transplant intervention including physical therapy, nutritional measures and psychological support scheduled for before the transplant may improve patient retention and compliance, better mitigate the effects of frailty and poor fitness after KT, and improve main outcomes in frail CKD patients.

The main objective is to assess effectiveness, feasibility and safety of a prehabilitation program (exercise, nutritional plans, psychological advice) in frail and non-frail KT candidates on clinical and functional outcomes after KT.

DETAILED DESCRIPTION:
Frailty is very frequent among patients with chronic kidney disease (CKD) included in the waiting list for deceased donor kidney transplantation (KT), and outcomes are worsened in those frail recipients after KT. Frailty and poor fitness powerfully predict mortality, kidney graft survival, and healthcareutilization after KT. Frailty in CKD patients displays a unique constellation of features such as muscle wasting, anorexia, protein energy wasting, inflammation, oxidative stress, catabolic/anabolic hormone imbalance, metabolic acidosis, and other cellularalterations that characterize a special population. Intervention is essential to improve quality of life for frail CKD patients, regardless of their age. Efforts to intervene with post- transplant physical therapy have been met with limited success, in large part due to high study dropout. A pre-transplant clinical framework for multimodal prehabilitation interventions including physicaltherapy, nutritional measures and psychological support scheduled for before the transplant may improve patient retention andcompliance, better mitigate the effects of frailty and poor fitness after KT, and improve main outcomes in frail CKD patients.

The main objective of this study is to assess effectiveness, feasibility and safety of multimodal prehabilitation (exercise, nutritional plans, psychological advice) in frail and non-frail KT candidates in the context of a randomized controlled clinical trial. The primary endpoint will be a composite achievement of clinical and functional outcomes in frail and non-frail KT candidates after KT.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with chronic kidney disease
* Inclusion in the waiting list for deceased donor kidney transplantation in the period September 2020 to August 2022

Exclusion Criteria:

* Patients unable to perform the exercise plan or giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bad-Outcome Composite Endpoint | 90 days post-kidney transplantation
  Delayed draft function >14 days + never functioning kidney + non-elective readmission before day 90 + surgical complications (wound healing problems, obstructive lymphocele, vascular thrombosis, urinary stenosis or leak, acute hemorrhage, immediate re-intervention) + discharge to an assisted facility + all-cause death.

SECONDARY OUTCOMES:
Changes in exercise capacity | Post-intervention (12 weeks)
  Changes in peak oxygen uptake (higher scores mean better outcome)
Changes in peripheral muscle strength | Post-intervention (12 weeks)
  Changes in handgrip and quadriceps muscles strength (higher scores mean better outcome)
Changes in respiratory muscle strength | Post-intervention (12 weeks)
  Changes in maximal inspiratory and expiratory muscle strength (higher scores mean better outcome)
Changes in physical activity | Post-intervention (12 weeks)
  Changes in physical activity assessed by activity monitors (higher scores mean better outcome)
Attendance | Post-intervention (12 weeks)
  Attended sessions (0-100%, patients are expected to attend a minimum of 80% sessions)
Exercise tolerability | Post-intervention (12 weeks)
  Patients not requiring exercise discontinuation or intensity modification
Changes in muscle mass | 1 month post-KT
  Changes in muscle mass assessed with total body dual energy X-ray
Changes in mood state | Through study completion, an average of 1 year
  Changes in Hospital Anxiety Depression Scale
Changes in health-related quality of life | Through study completion, an average of 1 year
  Score in the Short-Form 36 questionnaire (8 dimensions scoring 0-100, higher scores mean better outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Pascual Santos, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Saez MJ, Munoz-Redondo E, Morgado-Perez A, Delcros-Forestier L, Bach A, Faura A, Redondo D, Chamoun B, Burballa C, Buxeda A, Crespo M, Marco E, Pascual J; FRAILMar Study Group. Exercise-Based Prehabilitation for Kidney Transplant Candidates: the FRAILMar Randomized Controlled Trial. Am J Kidney Dis. 2025 Nov;86(5):634-645.e1. doi: 10.1053/j.ajkd.2025.07.003. Epub 2025 Aug 13. PMID 40816623
- [Derived] Perez-Saez MJ, Morgado-Perez A, Faura A, Munoz-Redondo E, Garriz M, Muns MD, Nogues X, Marco E, Pascual J. The FRAILMar Study Protocol: Frailty in Patients With Advanced Chronic Kidney Disease Awaiting Kidney Transplantation. A Randomized Clinical Trial of Multimodal Prehabilitation. Front Med (Lausanne). 2021 May 19;8:675049. doi: 10.3389/fmed.2021.675049. eCollection 2021. PMID 34095178